CLINICAL TRIAL: NCT01798485
Title: A Randomized, Phase 3 Study of Ganetespib in Combination With Docetaxel Versus Docetaxel Alone in Patients With Advanced Non-Small-Cell Lung Adenocarcinoma
Brief Title: A Phase 3 Study of Ganetespib in Combination With Docetaxel Versus Docetaxel Alone in Patients With Advanced NSCLC
Acronym: Galaxy 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped after the first Interim Analysis due to futility.
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9090-14; 2012-004349-34 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-25 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Non-Small-Cell Lung Adenocarcinoma; Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganetespib and Docetaxel (Experimental): Ganetespib (150 mg/m^2) and docetaxel (75 mg/m^2) were administered as separate 1-hour IV infusions on Day 1 of each 3-week treatment cycle. Administration of ganetespib preceded the administration of docetaxel. Ganetespib was administered again on Day 15 of each cycle.
  Interventions: Drug: Docetaxel; Drug: Ganetespib
- Docetaxel (Active Comparator): Docetaxel (75 mg/m^2) was administered on Day 1 of a 3-week treatment cycle by 1-hour IV infusion.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel, 75 mg/m^2, was administered according to prevailing practice and Investigator decision, generally until disease progression, intolerability, or patient's withdrawal of consent.
  Other Names: Taxotere; Docecad
Drug: Ganetespib — Ganetespib, 150 mg/m^2, was administered with docetaxel. After docetaxel treatment ceased, participants whose disease has not progressed continued to receive ganetespib alone until disease progression, unacceptable toxicity, or patient's withdrawal of consent.
  Other Names: STA-9090
  Arms: Ganetespib and Docetaxel

SUMMARY:
The purpose of this study is to determine whether combining ganetespib (STA-9090) with docetaxel is more effective than docetaxel alone in the treatment of patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Preliminary signals of clinical activity of ganetespib as a single agent have been observed in patients with advanced NSCLC. A Phase 2b/3 Study (9090-08) was initiated to evaluate the safety and activity of ganetespib in combination with docetaxel vs. docetaxel alone in NSCLC. Study 9090-08 is ongoing. Results from an interim analysis show that the combination has been well tolerated and an encouraging improvement in efficacy, including overall survival (OS) has been observed.

Update: An independent data monitoring committee (DMC) was established to review accumulating unblinded safety data, and efficacy data at two specified Interim Analyses. The DMC monitored the conduct of the trial (including the accrual/retention of patients) and reviewed the risks and benefits. The study was stopped after the first Interim Analysis due to futility.

The efficacy portion of this report is based on a 05 October 2015 data cut after the number of protocol-defined death events (336) for the first interim analysis had been achieved. The safety portion is based on the final database locked on 23 December 2015.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Stage IIIB or IV non-small-cell lung cancer (NSCLC)
* Eastern Oncology Cooperative Group (ECOG) Performance Status 0 or 1
* Prior therapy defined as 1 prior systemic therapy for advanced disease
* Documented disease progression during or following most first line therapy for advanced disease
* Adequate hematologic, hepatic, renal function

Exclusion Criteria:

* Epidermal growth factor receptor (EGFR) mutations
* Anaplastic lymphoma kinase (ALK) translocations
* Predominantly squamous, adenosquamous or unclear histologic type
* Active or untreated central nervous system (CNS) metastases
* Active malignancies other than NSCLC within the last 5 years with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin
* Serious cardiac illness or medical conditions
* Pregnant or lactating women
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (255):
- United States (76):
  - Arizona Oncology Associates PC- NAHOA, Flagstaff, Arizona
  - Arizona Oncology Associates, PC- NAHOA, Prescott Valley, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - City of Hope Comprehensive Breast Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - St. Joseph Hospital, Center for Cancer Prevention and Treatment, Orange, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - UC Davis Medical Center - UC Davis Comprehensive Cancer, Sacramento, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - City of Hope- South Pasadena, South Pasadena, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Eastern Connecticut Hematology Associates, Norwich, Connecticut
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Lynn Cancer Institute Center for Hematology Oncology, Boca Raton, Florida
  - Halifax Health - Medical Center, Daytona Beach, Florida
  - University of Miami Health System Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - University of South Florida - H. Lee Moffitt, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - University Of Chicago Medical Center, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc, Fort Wayne, Indiana
  - AAMC Oncology and Hematology, Annapolis, Maryland
  - The Center for Cancer and Blood Disorders (CCBD) - Bethesda, Bethesda, Maryland
  - The John R Marsh Cancer Center, Hagerstown, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Luke's Hospital Duluth, Duluth, Minnesota
  - Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - St. Louis Cancer Care, LLP - North County, Bridgeton, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Clinical Research Alliance, Lake Success, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - New Hanover Regional Medical Center - Zimmer Cancer Center, Wilmington, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Tulsa Cancer Institute, PLLC, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Prairie Lakes Healthcare System, Watertown, South Dakota
  - Erlanger Institute for Clinical Research, Chattanooga, Tennessee
  - Associates In Oncology and Hematology, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Oncology-Arlington North, Arlington, Texas
  - Texas Oncology - Arlington South, Arlington, Texas
  - Texas Oncology, P.A., Beaumont, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Simmons Comprehensive Cancer Center, Dallas, Texas
  - Houston Methodist Hospital Research Institute, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cancer Care Centers Of South Texas, San Antonio, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Providence Regional Medical Center Everett, Everett, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Mary Babb Cancer Center, Morgantown, West Virginia
  - Green Bay Oncology, Ltd. - St. Mary's Site, Green Bay, Wisconsin
  - Green Bay Oncology, Green Bay, Wisconsin
- Austria (8):
  - Landesklinikum Krems, Krems, Lower Austria
  - Bezirkskrankenhaus Kufstein [Onkologie], Kufstein, Tyrol
  - Krankenhaus Der Barmherzigen Schwestern, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Allgemeines Krankenhaus Linz, Linz
  - Elisabeth Linz Hospital, Linz
  - Otto Wagner Spital, Vienna
  - Sozialmedizinisches Zentrum Baumgartner Höhe, Vienna
- Belgium (8):
  - AZ Sint-Maarten - Campus Leopoldstraat, Mechelen, Antwerpen
  - Clinique Saint-Pierre Ottignies, Ottignies, Brabant Wallon
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi, Hainaut
  - INDC Entité Jolimontoise - Polyclinique de Jolimont, Haine-Saint-Paul, Hainaut
  - CHU Dinant Godinne UCL Namur, Yvoir, Namur
  - Algemeen Stedelijk Ziekenhuis - Campus Aalst, Roeselaere, West-Vlaanderen
  - Cliniques Universitaire Saint-Luc, Brussels
  - CHR de la Citadelle - Site Citadelle, Liège
- Bosnia and Herzegovina (7):
  - Clinical Centre Banja Luka, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla, Tuzla, Tuzlanski kanton
  - Clinical Hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Clinic of Oncology, Sarajevo
  - University Clinical Centre Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
  - Kantonalna bolnica Zenica, Zenica
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Mc Gill University-MUHC, Montreal, Quebec
- Croatia (2):
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Opca bolnica Pula, Pula, Istria County
- Czechia (4):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Na Bulovce, Prague
- France (10):
  - CHI des Alpes du Sud, Gap, Hautes-Alpes
  - Centre D'Oncologie Du Pays Basque, Bayonne, Pyrénées-Atlantiques
  - Centre Hosptalier De Villefranche-Sur-Saone, Villefranche-sur-Saône, Rhône
  - Chi creteil, Créteil, Val-de-Marne
  - Chu De Grenoble - Hopital Michallon, Grenoble
  - Centre Léon Bérard, Lyon
  - Groupe Hospitalier Cochin, Paris
  - Centre Hospitalier Universitaire de Rennes - Hopital d, Rennes
  - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg, Strasbourg
- Germany (21):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universiaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen, Baden-Wurttemberg
  - Asklepios Fachklinik München-Gauting, Gauting, Bavaria
  - Klinikum Bogenhausen, Munich, Bavaria
  - Gesundheitszentrum Wetterau, Bad Nauheim, Hesse
  - Johann Wolfgang Goethe University Clinic Frankfurt, Frankfurt am Main, Hesse
  - Klinikum Kassel, Kassel, Hesse
  - Kliniken der Stadt Köln gGmbH, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Leipzig [Pneumologie], Leipzig, Saxony
  - Pneumologisches Forschungsinstitut an der Lungenclinic Gross, Großhansdorf, Schleswig-Holstein
  - MVZ Äerzteforum Seestraße, Berlin
  - Ev. Krankenhaus Bielefeld, Bielefeld
  - Klinikum Frankfurt An Der Oder, Frankfurt (Oder)
  - Practice Laack, Hamburg
  - Unikl. Schleswig-Holstein - Lübeck, Lübeck
  - J. Gutenberg Uni.Mainz, Mainz
  - Medizinische Fakultät Mannheim Uni Heidelberg, Mannheim
  - Gemeinschaftspraxis fuer Haematologie und Onkologie, Münster
  - Klinikum Offenbach GmbH, Offenbach
- Hungary (7):
  - Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkó, Deszk, Csongrád megye
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár, Fejér
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest, Pest County
  - Semmelweis Egyetem, Budapest
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Békés Megyei Pándy Kálmán Kórház, Gyula
  - CRU Hungary Kft., Miskolc
- Italy (13):
  - Irccs Irst, Meldola, Forli
  - Presidio Ospedaliero Centrale Belcolle, AUSL Viterbo, Viterbo, Lazio
  - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - CRO, IRCCS, Istituto Nazionale Tumori, Aviano, Pordenone
  - Istituti Fisioterapici Ospitalieri Regina Elena, Roma, Roma
  - Azienda Policlinico Umberto I, Rome, Roma
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - AOU S.Martino, IRCCS, IST-Istituto Nazionale Ricerca Sul Can, Genova
  - Istituto Europeo di Oncologia, Istituto di Ricovero e Cura a, Milan
  - Iov-Irccs, Padua
  - Ospedale S.Maria della Misericordia, AO di Perugia, Universi, Perugia
  - Ospedale Guglielmo da Saliceto, AUSL Piacenza, Piacenza
  - Borgo Roma, Policlinico G.Rossi, AOU Integrata Verona, Verona
- Netherlands (6):
  - Ziekenhuis Assen, Assen, Drenthe
  - Ziekenhuis St Jansdal, Harderwijk, Gelderland
  - Gelre Ziekenhuis Zutphen, Zutphen, Gelderland
  - academisch ziekenhuis Maastricht, Maastricht, Limburg
  - Isala Klinieken Zwolle, Zwolle, Overijssel
  - Sint Antoniusziekenhuis, location Utrecht, Utrecht
- Poland (12):
  - NZOZ Med Polonia, Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan, Greater Poland Voivodeship
  - Medica Pro Familia Sp. z o.o. S.K.A., Krakow, Lesser Poland Voivodeship
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock, Masovian Voivodeship
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej - Curie, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Szpital Wojewodzki w Lomzy im. Kardynala S. Wyszynskiego, Łomża, Podlaskie Voivodeship
  - Szpital Wojewodzki Zespolony, Elblag, Warmian-Masurian Voivodeship
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Szpital Chorob Pluc im. Sw. Jozefa w Pilchowicach, Pilchowice
  - Szpital Specjalistyczny, Prabuty
  - Wojewodzki Szpital Specjalistyczny im. M.Kopernika, Lodz, Łódź Voivodeship
- Romania (8):
  - Institutul Oncologic "Prof. Dr. Alex. Trestioreanu", Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Oncologic "Prof.Dr.I.Chiricuta" Cluj Napoca, Cluj-Napoca
  - Medisprof, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Oncomed, Timișoara
- Russia (20):
  - Synta Pharmaceuticals Investigational Site, Chelyabinsk
  - Synta Pharmaceuticals Investigational Site, Ivanovo
  - Synta Pharmaceuticals Investigational Site, Izhevsk
  - Synta Pharmaceuticals Investigational Site, Kemerovo
  - Synta Pharmaceuticals Investigational Site, Krasnoyarsk
  - Synta Pharmaceuticals Investigational Site, Kursk
  - Synta Pharmaceuticals Investigational Site, Lipetsk
  - Synta Pharmaceuticals Investigational Site, Moscow
  - Synta Pharmaceuticals Investigational Site, Nizhny Novgorod
  - Synta Pharmaceuticals Investigational Site, Novosibirsk
  - Synta Pharmaceuticals Investigational Site, Omsk
  - Synta Pharmaceuticals Investigational Site, Oryol
  - Synta Pharmaceuticals Investigational Site, Rostov-on-Don
  - Synta Pharmaceuticals Investigational Site, Saint Petersburg
  - Synta Pharmaceuticals Investigational Site, Samara
  - Synta Pharmaceuticals Investigational Site, Saransk
  - Synta Pharmaceuticals Investigational Site, Sochi
  - Synta Pharmaceuticals Investigational Site, Stavropol
  - Synta Pharmaceuticals Investigational Site, Ufa
  - Synta Pharmaceuticals Investigational Site, Yekaterinburg
- Serbia (5):
  - Clinical Centre of Serbia, Belgrade, Belgrade
  - Clinical Centre Nis, Niš, Nišavski okrug
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Institute for pulmonary diseases of Vojvodine, Kamenitz
  - Clinical Center Kragujevac, Kragujevac, Šumadijski okrug
- Slovenia (2):
  - Univerzitetna klinika za pljucne bolesti in alergijo Golnik, Golnik
  - Onkoloski institut Ljubljana, Ljubljana
- Spain (18):
  - Xerencia de Xestión Integrada A Coruña Hospital Teresa Herrera, A Coruña, A Coruña
  - Synta Pharmaceuticals Investigational Site, Málaga, Andalusia
  - H. Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital de Mataró, Consorci Sanitari del Maresme, Mataró, Barcelona
  - Synta Pharmaceuticals Investigational Site, Santander, Cantabria
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Synta Pharmaceuticals Investigational Site, Oviedo, Principality of Asturias
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - H.U. Vall d'Hebrón, Barcelona
  - Synta Pharmaceuticals Investigational Site, Barcelona
  - H.U. Reina Sofía, Córdoba
  - Synta Pharmaceuticals Investigational Site, Girona
  - Synta Pharmaceuticals Investigational Site, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - F. Jiménez Diaz, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Ukraine (16):
  - Synta Pharmaceuticals Investigational Site, Cherkasy
  - Synta Pharmaceuticals Investigational Site, Chernivtsi
  - Synta Pharmaceuticals Investigational Site, Dnipro
  - Synta Pharmaceuticals Investigational Site, Donetsk
  - Synta Pharmaceuticals Investigational Site, Ivano-Frankivsk
  - Synta Pharmaceuticals Investigative Site, Kharkiv
  - Synta Pharmaceuticals Investigational Site, Khmelnytskyi
  - Synta Pharmaceuticals Investigational Site, Kirovohrad
  - Synta Pharmaceuticals Investigational Site, Kryvyi Rih
  - Synta Pharmaceuticals Investigational Site, Kyiv
  - Synta Pharmaceuticals Investigational Site, Makiivka
  - Synta Pharmaceuticals Investigational Site, Poltava
  - Synta Pharmaceuticals Investigational Site, Simferopol
  - Synta Pharmaceuticals Investigational Site, Sumy
  - Synta Pharmaceuticals Investigational Site, Uzhhorod
  - Synta Pharmaceuticals Investigational Site, Vinnytsia
- United Kingdom (10):
  - Synta Pharmaceuticals Investigational Site, Truro, Cornwall
  - Synta Pharmaceuticals Investigational Site, Shrewsbury, Shropshire
  - Synta Pharmaceuticals Investigational Site, Sutton, Surrey
  - Synta Pharmaceuticals Investigational Site, Swindon, Wiltshire
  - Synta Pharmaceuticals Investigational Site, Cardiff
  - Synta Pharmaceuticals Investigational Site, Edinburgh
  - Synta Pharmaceuticals Investigational Site, Leicester
  - Synta Pharmaceuticals Investigational Site, London
  - Synta Pharmaceuticals Investigational Site, Nottingham
  - Synta Pharmaceuticals Investigational Site, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 209 sites screened at least one patient and 175 sites randomized at least one patient.
Pre-assignment Details: 1220 patients with advanced NSCLC of adenocarcinoma histology diagnosed ≥6 months prior to study entry were screened. 696 patients were randomized in a 1:1 ratio to two arms and stratified by:
  * ECOG (0 versus 1)
  * Screening total LDH levels (normal vs. elevated)
  * Geographic region (North America and Western Europe vs. Rest of World)
Period: Overall Study
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Started | 347 | 349
Safety Population as of 23 Dec 2015 | 338 | 342
Randomized as of 19 October 2015 | 335 | 337
Completed | 1 | 59
Not Completed | 346 | 290
Not completed — Adverse Event | 32 | 40
Not completed — Withdrawal by Subject | 27 | 31
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 14 | 10
Not completed — Objective Disease Progression | 152 | 106
Not completed — Death | 25 | 22
Not completed — Sponsor Decision | 61 | 54
Not completed — Clinical Progression | 35 | 24

BASELINE CHARACTERISTICS:
Population: All randomized participants as of 23 December 2015
Groups:
- Total: Total of all reporting groups
Arm/Group | Ganetespib and Docetaxel | Docetaxel | Total
Number analyzed (Participants) | 347 | 349 | 696
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.93) | 60.1 (8.69) | 60.5 (8.81)
Age, Customized [Number; unit: participants]
  <65 years | 227 | 247 | 474
  >=65 years | 120 | 102 | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 135 | 276
  Male | 206 | 214 | 420
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 341 | 340 | 681
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Geographic region [Number; unit: participants]
  North America | 41 | 44 | 85
  Western Europe | 101 | 96 | 197
  Rest of World | 205 | 209 | 414
Smoking History [Number; unit: participants]
  Never Smoked | 62 | 62 | 124
  Ever Smoked | 282 | 284 | 566
  Unknown | 3 | 3 | 6
Time from Advanced NCSLC Diagnosis to Consent [Mean (Standard Deviation); unit: months] — NCSLC = non-small-cell lung cancer
  months | 11.54 (5.995) | 11.76 (7.740) | 11.65 (6.920)
Stage at Initial Diagnosis [Number; unit: participants] — Disease stage described using American Joint Committee on Cancer (AJCC). Stages ranged from I (cancer was small and had not spread to the lymph nodes) to IV (cancer spread throughout the body). Stage III (cancer had spread to nearby tissue or lymph nodes) was further differentiated based on regional lymph nodes: Stage IIIA (spread to nearby lymph nodes) and Stage IIIB (spread to distance lymph nodes).
  participants
    I/II | 22 | 19 | 41
    IIIA | 18 | 18 | 36
    IIIB | 52 | 52 | 104
    IV | 254 | 258 | 512
    Unknown | 1 | 2 | 3
ECOG at Study Entry [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants' disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  participants
    0 = Fully Active | 124 | 125 | 249
    1 = Restrictive but Ambulatory | 223 | 224 | 447
    2 = Ambulatory unable to Work | 0 | 0 | 0
    3 = Limited Self-Care | 0 | 0 | 0
    4 = Completely Disabled | 0 | 0 | 0
Lactate Dehydrogenase (LDH) at Study Entry [Number; unit: participants]
  Normal | 246 | 247 | 493
  Elevated | 101 | 102 | 203
Brain Metastasis [Number; unit: participants]
  Yes | 65 | 55 | 120
  No | 282 | 294 | 576
Bone Metastasis [Number; unit: participants]
  Yes | 115 | 100 | 215
  No | 232 | 249 | 481
Intra-Thoracic Metastasis only [Number; unit: participants]
  Yes | 95 | 120 | 215
  No | 252 | 229 | 481

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival as of 19 October 2015
Description: Overall survival (OS) was measured from the date of randomization to the date of death from any cause.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
months | 10.9 [9.0 to 12.3] | 10.5 [8.6 to 12.2]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Primary study hypothesis was tested at a 2-sided, 0.05 significance level using a stratified log-rank test; Test type: Superiority or Other; p = 0.3293, Log Rank; P-value was from stratified log-rank test (strata: screening LDH, screening ECOG and geographic region); Hazard Ratio (HR) = 1.111, 95% CI 2-sided [0.899 to 1.372]
Statistical Analysis 2: Comparison: Ganetespib and Docetaxel vs Docetaxel; Futility analysis for the first Interim Analysis which had a database cutoff of 19 October 2015. For the first interim analysis, if the lower limit of the 2-sided 99.5% confidence interval (CI) for the Hazard Ratio was greater than 0.75, then the study could be stopped for futility, based on Data Monitoring Committee recommendation. Hazard ratio and 99.5% CI were calculated using the stratified Cox Proportional Hazards model (strata: screening LDH, screening ECOG and geographic region); Test type: Superiority or Other; Hazard Ratio (HR) = 1.111, 99.5% CI 2-sided [0.821 to 1.503]

2. Secondary Outcome: Progression-free Survival (PFS) as of 19 October 2015
Description: The progression-free interval is the interval from the date of randomization until tumor progression per modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1), clinical progression, or death from any cause in the absence of progressive disease, whichever occurs first. Data represents the investigator's assessment.
  Progressive Disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
months | 4.2 [3.8 to 4.4] | 4.3 [3.6 to 5.6]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.1180, Log Rank — Significance level of 0.05; Stratified log-rank test with stratification variables, ECOG, screening total LDH levels, and geographic region, used to compare the treatment groups; Hazard Ratio (HR) = 1.161, 95% CI 2-sided [0.961 to 1.403]

3. Secondary Outcome: Overall Survival (OS) In Participants With an Elevated Screening Lactate Dehydrogenase (eLDH) as of 19 October 2015
Description: OS was measured from the date of randomization to the date of death from any cause. Elevated LDH includes values above the upper limit of normal.
Time Frame: up to 36 months
Population: Randomized participants with elevated LDH at screening
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 99 | 98
months | 7.1 [5.4 to 11.0] | 9.0 [6.2 to 10.3]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.2506, Log Rank — Significance level of 0.05; P-value was from stratified log-rank test (strata: screening ECOG and geographic region); Hazard Ratio (HR) = 1.232, 95% CI 2-sided [0.865 to 1.754]

4. Secondary Outcome: Objective Response Rate (ORR) as of 19 October 2015
Description: Percentage of participants whose best overall response, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), was either a complete response (CR) or a partial response (PR).
  CR was defined as the disappearance (or normalization) of all target lesions. PR was defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
percentage of participants | 13.7 [10.2 to 17.9] | 16.0 [12.3 to 20.4]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.448, Fisher Exact — Significance level of 0.05

5. Secondary Outcome: Disease Control Rate (DCR) as of 19 October 2015
Description: Percentage of participants whose best overall response, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), was either a complete response (CR), a partial response (PR), or stable disease (SD).
  CR was defined as the disappearance (or normalization) of all target lesions. PR was defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study. For participants with a best response of SD, duration of SD must be for at least 6 weeks or 12 weeks.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
percentage of participants
  >=6 weeks | 64.9 [59.1 to 69.6] | 60.8 [55.4 to 66.1]
  >=12 weeks | 46.0 [40.5 to 51.5] | 46.9 [41.5 to 52.4]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; >= 6 weeks; Test type: Superiority or Other; p = 0.339, Fisher Exact — Significance level of 0.05
Statistical Analysis 2: Comparison: Ganetespib and Docetaxel vs Docetaxel; >= 12 weeks; Test type: Superiority or Other; p = 0.817, Fisher Exact — Significance level of 0.05

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) as of 19 October 2015
Description: Only participants who achieved a confirmed response (complete response (CR) or partial response (PR)) were included in the DOR analysis.
  CR was defined as the disappearance (or normalization) of all target lesions.
  PR was defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
Time Frame: up to 36 months
Population: Randomized participants who had a confirmed response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 46 | 54
months | 5.8 [3.0 to 5.9] | 5.8 [4.3 to 6.9]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.0111, Log Rank — Significance level of 0.05; P-value was from stratified log-rank test (strata: screening LDH, screening ECOG and geographic region); Hazard Ratio (HR) = 2.344, 95% CI 2-sided [1.207 to 4.551]

7. Secondary Outcome: Progression Free Survival (PFS) in Participants With an Elevated Screening Lactate Dehydrogenase (eLDH) as of 19 October 2015
Description: The progression-free interval is the interval from the date of randomization until tumor progression per modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1), clinical progression, or death from any cause in the absence of progressive disease, whichever occurs first. Data represents the investigator's assessment.
  Progressive Disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Elevated LDH includes values above the upper limit of normal.
Time Frame: up to 36 months
Population: Randomized participants who had an elevated screening LDH
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 99 | 98
months | 3.0 [2.4 to 4.0] | 2.8 [2.2 to 4.1]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.5191, Log Rank — Significance level of 0.05; P-value was from stratified log-rank test (strata: screening ECOG and geographic region); Hazard Ratio (HR) = 1.112, 95% CI 2-sided [0.797 to 1.551]

8. Secondary Outcome: Objective Response Rate (ORR) in Participants With an Elevated Screening Lactate Dehydrogenase (eLDH) as of 19 October 2015
Description: Percentage of participants whose best overall response, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), was either a complete response (CR) or a partial response (PR).
  CR was defined as the disappearance (or normalization) of all target lesions.
  PR was defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  Elevated LDH includes values above the upper limit of normal.
  This study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Time Frame: up to 36 months
Population: Randomized participants who had an elevated screening LDH. However, this study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Disease Control Rate (DCR) in Participants With an Elevated Screening Lactate Dehydrogenase (eLDH) as of 19 October 2015
Description: Percentage of participants whose best overall response, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), was a complete response (CR), a partial response (PR), or stable disease (SD).
  CR was defined as the disappearance (or normalization) of all target lesions.
  PR was defined as <=30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study. The duration of SD must be for at least 6 weeks or 12 weeks.
  Elevated LDH includes values above the upper limit of normal.
  This study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Time Frame: up to 36 months
Population: as for outcome 8
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Kaplan-Meier Estimate for Time to Emergence of New Metastatic Lesion (TNL) as of 19 October 2015
Description: TNL was defined as time from the randomization date to the first day of radiological progression that included new metastatic lesions. Participants with no new metastatic lesions were censored at the date of the most recent radiological assessment.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
months | 8.1 [6.5 to 9.7] | 8.7 [7.2 to 11.6]
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.1343, Log Rank — Significance level of 0.05; Stratified log-rank test (strata: screening LDH, screening ECOG and geographic region); Hazard Ratio (HR) = 1.233, 95% CI 2-sided [0.937 to 1.621]

11. Secondary Outcome: Percentage of Participants With Progressive Disease Due to Any New Metastatic Lesion as of 19 October 2015
Description: Progressive disease was due to either new metastatic lesions only or new metastatic lesions and target tumor growth.
Time Frame: up to 36 months
Population: Randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 335 | 337
percentage of participants | 34.9 | 30.6
Statistical Analysis 1: Comparison: Ganetespib and Docetaxel vs Docetaxel; Test type: Superiority or Other; p = 0.250, Fisher Exact — Significance level of 0.05

12. Other Pre Specified Outcome: Exploratory Biomarker Analyses
Description: Exploratory biomarker analyses was to assess correlation between biomarkers and clinical outcome. However, this study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Time Frame: up to 36 months
Population: Randomized
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Participants With Treatment-Emergent Adverse Events as of 23 December 2015
Description: Treatment-emergent adverse events (AEs) were defined as AEs that occurred from the time of first dose through 30 days after the last dose of study medication. The Investigator graded the severity of AEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria:
  Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death A Serious AE (SAE) is defined as any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or constitutes an important medical event.
Time Frame: up to 36 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 338 | 342
participants
  >=1 AE | 317 | 307
  >=1 AE with CTCAE grade of 3 or 4 | 222 | 184
  >=1 SAE | 139 | 107
  >=1 AE leading to dose reduction | 61 | 37
  >=1 AE leading to delayed dose | 125 | 55
  >=1 AE leading to study drug discontinuation | 31 | 36
  >=1 SAE leading to study drug discontinuation | 19 | 15
  >=1 SAE leading to hospitalization | 109 | 87
  >=1 SAE with outcome of death | 40 | 30
  >=1 AE with first occurrence during Cycle 1-2 | 280 | 280
  >=1 AE with first occurrence during Cycle 1-4 | 304 | 299
  >=1 AE with first occurrence during Cycle 1-6 | 312 | 302

14. Secondary Outcome: Patient-Reported Quality of Life as Measured by the European Quality Of Life - Five Dimensions - Three Levels (EQ-5D-3L) Survey
Description: The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. An overall EQ-5D-3L index was calculated (see EuroQoL website, http://www.euroqol.org/eq-5d-products/eq-5d-3l.html), with an index of 1.0 representing full health and and "0" represents dead, with some health states being worse than dead (<"0").
  This study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Time Frame: Day 1 (pre-treatment), Day 63 (Cycle 3 Day 1), Day 105 (Cycle 5 Day 1) and end of trial
Population: Randomized participants. However, this study stopped prematurely due to futility and development of this product ceased. The sponsor made a decision at that time to not analyze this outcome. The sponsor no longer has staff or capabilities for further analysis.
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Patient-Reported Symptom Improvement as Measured by the Functional Assessment of Cancer Therapy - Lung (FACT-L) Version 4 Test
Description: The FACT-L contains 4 general subscales and a Lung Cancer Subscale (LCS). General subscales include: Physical Well-Being (PWB), Social/ Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). The LCS assesses symptoms commonly reported by lung cancer patients (e.g., shortness of breath, weight loss, and tightness in the chest). The FACT-L total score ranges from 0 to 136, higher scores represent better QOL.
  Data were not summarized due to the early termination of the study due to futility.
Time Frame: Day 1 (pre-treatment), Day 63 (Cycle 3 Day 1), Day 105 (Cycle 5 Day 1) and end of trial
Population: Randomized participants
Arm/Group | Ganetespib and Docetaxel | Docetaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 36 months
Arm/Group | Docetaxel | Ganetespib and Docetaxel
Serious Adverse Events (participants affected / at risk) | 107/342 | 139/338
Other Adverse Events (participants affected / at risk) | 293/342 | 308/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=342) | Ganetespib and Docetaxel (N=338)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11) | 19 (20)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 10 (15) | 12 (14)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 15 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3)
Asthenia (General disorders) | 1 (1) | 7 (9)
Chest pain (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2) — When an SAE of death is received, the site is queried to request additional information. If the site is not able to determine a specific adverse event, they report 'death' as the event.
Fatigue (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 5 (6)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 3 (3) | 0 (0)
Sudden death (General disorders) | 0 (0) | 3 (3)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Immunodeficiency (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 5 (5)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 12 (12)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Investigations) | 0 (0) | 2 (2)
Hypovolaemia (Investigations) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 16 (16)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 4 (4)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=342) | Ganetespib and Docetaxel (N=338)
Anaemia (Blood and lymphatic system disorders) | 70 (144) | 59 (106)
Leukopenia (Blood and lymphatic system disorders) | 18 (54) | 20 (39)
Neutropenia (Blood and lymphatic system disorders) | 94 (255) | 109 (243)
Constipation (Gastrointestinal disorders) | 26 (31) | 35 (41)
Diarrhoea (Gastrointestinal disorders) | 47 (64) | 149 (327)
Nausea (Gastrointestinal disorders) | 68 (103) | 59 (86)
Stomatitis (Gastrointestinal disorders) | 36 (52) | 32 (40)
Vomiting (Gastrointestinal disorders) | 23 (27) | 36 (46)
Asthenia (General disorders) | 48 (109) | 51 (100)
Chest pain (General disorders) | 17 (20) | 19 (26)
Fatigue (General disorders) | 72 (123) | 79 (130)
Oedema peripheral (General disorders) | 29 (30) | 28 (39)
Pyrexia (General disorders) | 19 (30) | 26 (33)
Infusion related reaction (Injury, poisoning and procedural complications) | 11 (13) | 17 (32)
Weight decreased (Investigations) | 18 (22) | 38 (50)
Decreased appetite (Metabolism and nutrition disorders) | 35 (49) | 52 (66)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (20) | 26 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (35) | 17 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (19) | 24 (28)
Bone pain (Musculoskeletal and connective tissue disorders) | 17 (24) | 19 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (52) | 38 (64)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (19) | 18 (23)
Dizziness (Nervous system disorders) | 21 (30) | 24 (41)
Headache (Nervous system disorders) | 17 (23) | 22 (30)
Neuropathy peripheral (Nervous system disorders) | 33 (52) | 41 (63)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (29) | 15 (18)
Insomnia (Psychiatric disorders) | 8 (8) | 23 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 34 (45)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (56) | 55 (59)
Alopecia (Skin and subcutaneous tissue disorders) | 84 (98) | 76 (93)
Rash (Skin and subcutaneous tissue disorders) | 16 (20) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right, 60 days before submission for publication, to review disclosures and require deletion of its confidential information, excluding the study results. Public disclosure shall be delayed for up to 60 additional days in order for the Sponsor to file a patent application, if needed. Single center publications will be postponed until after disclosure of pooled data (all sites), or, for a period of 18 months from study completion/termination at all participating sites.